CLINICAL TRIAL: NCT04640142
Title: Prospective, Open-label, Single-arm, Multicentre Phase 3 Study to Evaluate the Pharmacokinetics, Efficacy, Tolerability, and Safety of Subcutaneous Human Immunoglobulin (Newnorm) in Patients With Primary Immunodeficiency Diseases
Brief Title: Study to Evaluate the Pharmacokinetics, Efficacy, Tolerability, and Safety of Subcutaneous Human Immunoglobulin (Newnorm) in Patients With Primary Immunodeficiency Diseases
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NORM-01
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Primary Immune Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Newnorm (Experimental): Newnorm is a 20% human normal immunoglobulin for SC infusion
  Interventions: Biological: Newnorm

INTERVENTIONS:
Biological: Newnorm — Newnorm is a 20% human normal immunoglobulin for SC infusion.

SUMMARY:
Prospective, open-label, single-arm, multicentre Phase 3 study to evaluate the pharmacokinetics, efficacy, tolerability, and safety of subcutaneous human immunoglobulin (Newnorm) in patients with primary immunodeficiency diseases

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥2 years and ≤75 years
2. Documented and confirmed diagnosis of PID as defined by European Society of Immunodeficiencies (ESID) and the Pan American Group for Immune Deficiency (PAGID) and requiring immunoglobulin replacement therapy due to hypogammaglobulinaemia or agammaglobulinaemia. The exact type of PID must be recorded.
3. At least 12 weeks of regular treatment before the screening visit (i.e., with a stable dosing interval) with any IVIG, SCIG, or fSCIG, with a stable IgG dose between 200 and 800 mg/kg/month. A stable dose is defined as one that deviates less than ±25% from the mean dose for all infusions within this 12-week period before screening.
4. Trough level of IgG ≥5 g/L at screening and documentation of an IgG trough level of ≥5 g/L at least once within the previous 12 weeks.
5. Freely given written informed consent from adult patients or freely given written informed consent from the patient's parent(s)/legal guardian(s) and written informed assent from paediatric or adolescent patients in accordance with the applicable regulatory requirements, before any study-specific procedure takes place.
6. Willingness to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

Exclusion Criteria:

1. Any acute infection requiring IV antibiotic treatment within 2 weeks before the screening visit or during the screening period, or any SBI within the 3 months prior to the screening visit or during the screening period.
2. The patient has isolated specific antibody deficiency disorder, isolated IgG subclass deficiency, or transient hypogammaglobulinaemia of infancy.
3. Current medical condition or history of condition known to cause secondary immune deficiency, for example, chronic lymphocytic leukaemia, lymphoma, multiple myeloma, or chronic or recurrent neutropenia (absolute neutrophil count <1000/μL).
4. Known history of ADRs to IgA contained in other products.
5. Body mass index >40 kg/m2.
6. Exposure to blood or any blood product or plasma derivative other than IgG for PID within 3 months before the first infusion of Newnorm.
7. History of or ongoing severe hypersensitivity, e.g., anaphylaxis or severe systemic response, or persistent reactions to blood or plasma-derived products, or to any component of Newnorm (such as glycine).
8. Severe liver dysfunction (alanine aminotransferase [ALT] >3 times the upper limit of normal for the expected normal range for the testing laboratory) at screening.
9. Known protein-losing enteropathies or proteinuria (known urinary protein loss of >1 g/24 h, or dipstick proteinuria of ≥3+).
10. Moderate to severe renal dysfunction (per investigator discretion based on estimated glomerular filtration rate [eGFR] ≤44 mL/min/1.73 m2, as defined by KDIGO Clinical Practice Guideline) or predisposition to acute renal failure (e.g., any degree of pre-existing renal dysfunction in presence of additional acute renal failure risk factors, e.g. routine treatment with known nephrotoxic drugs).
11. Uncontrolled diabetes mellitus (HbA1c > 7% / >53 mmol/mol).
12. Uncontrolled arterial hypertension (systolic blood pressure of ≥ 130 mmHg for the subject under 13 years of age, ≥ 140 mmHg for subject 13 to 17 years of age, and > 160 mmHg for adults).
13. Dysrhythmia/Tachycardia (resting heart rate > 100 bpm for adults/adolescents and > 120 bpm for children) and symptomatic bradycardia (resting heart rate < 60 bpm for adults, < 50 bpm for adolescents, and < 75 bpm for children in presence of symptoms e.g., low blood pressure, abnormal rhythm, chest discomfort, shortness of breath). Physiological sinus bradycardia in physically active adults/children/athletes is NOT an exclusion criterion).
14. The subject has a history of or current diagnosis of deep venous thrombosis or thromboembolism (e.g. myocardial infarction, cerebrovascular accident, or transient ischemic attack); history refers to an incident in the year prior to screening or 2 episodes over lifetime.
15. The subject is currently receiving anti-coagulation therapy which would make SC administration inadvisable (vitamin K antagonist, nonvitamin K antagonist oral anticoagulants [e.g. dabigatran etexilate targeting Factor IIa, rivaroxaban, edoxaban, and apixaban targeting Factor Xa], parenteral anticoagulants [e.g. fondaparinux]).
16. Treatment with oral or parenteral steroids either

    1. at daily doses >0.3 mg/kg of prednisone (or equivalent) within the last 12 weeks before screening or
    2. bolus treatment of a daily dose greater than 1 mg/kg of prednisone (or equivalent) for longer than 10 days within the last 12 weeks before screening. Courses of corticosteroids (intermittent) of not more than 10 days would not exclude a patient. Inhaled or topical corticosteroids are allowed.
17. Treatment with systemic immunosuppressants including chemotherapeutic agents 1 year before screening or immunomodulatory drugs 12 weeks before the screening visit.
18. Live viral vaccination (such as measles, rubella, mumps, or varicella) within 1 month before the first infusion of Newnorm, during the study period, and within 3 months after last infusion of Newnorm. Note: Seasonal inactivated (killed) influenza vaccines (incl. H1N1) are allowed. COVID vaccines (mRNA vaccine and a non-replicating viral vector vaccine) are allowed.
19. Treatment with any investigational medicinal product (IMP) within 3 months before the screening visit.
20. Presence of any condition likely to interfere with the evaluation of Newnorm or with the compliant conduct of the study.
21. Known or suspected abuse of alcohol, drugs, and/or psychotropic agents within 12 months before screening.
22. Known human immunodeficiency virus (HIV)-1/2, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection or positive for HIV-1/2, HBV, or HCV at screening.
23. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to use an effective birth control method (refer to protocol Section 7.4.10.b) while on study and for 30 days following the last dose of study drug.
24. Men who are unwilling to use birth control to prevent pregnancy for the duration of the study (unless the female partner

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Bacterial Infections | 52 weeks
  Rate of SBIs (defined as bacteraemia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, and visceral abscess) per person-year on treatment.
Average total IgG concentration | 16 weeks
  Average total IgG concentration (Cav) on steadystate dosing.

SECONDARY OUTCOMES:
Infections of any type of seriousness | 52 weeks
  Infections of any type or seriousness (including acute sinusitis, exacerbation of chronic sinusitis, acute otitis media, acute bronchitis, infectious diarrhoea, etc) (total and by category, annual rate)
Time to resolution of infections | 52 weeks
  Time to resolution of infections
Use of antibiotics | 52 weeks
  Use of antibiotics (number of days on antibiotics and annual rate of treatment episodes) characterised as therapeutic or prophylactic use
Hospitalisations due to infection | 52 weeks
  Hospitalisations due to infection (number of days and annual rate)
Episodes of fever | 52 weeks
  Episodes of fever
Days lost from work, school, kindergarten, or day care due to infection | 52 weeks
  Days lost from work, school, kindergarten, or day care due to infection
Child Health Questionnaire-Parent Form | 52 weeks
  Child Health Questionnaire-Parent Form (CHQPF50) for patients <14 years
SF-36 Health Survey | 52 weeks
  SF-36 Health Survey for patients ≥ 14 of age
Non-compartmental PK analyses of all available PK profiles (IVIG and SCIG) | 16 weeks
  Total IgG, IgG subclasses (IgG1, IgG2, IgG3, and IgG4), and antigen specific antibodies against Haemophilus influenzae B (capsular polysaccharide), Streptococcus pneumoniae (serotypes 4, 6B, 9V, 14, 18C, 19F, 23F), cytomegalovirus (CMV), tetanus, and measles
IgG Levels | 16 weeks
  Trough and peak levels of total IgG and IgG subclasses for weekly Newnorm relative to 3- or 4-weekly IVIG dosing

CONTACTS AND LOCATIONS:
Locations (22):
- United States (11):
  - Octapharma Research Site, Irvine, California
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, Hollywood, Florida
  - Octapharma Research Site, Port Saint Lucie, Florida
  - Octapharma Research Site, St. Petersburg, Florida
  - Octapharma Research Site, Chicago, Illinois
  - Octapharma Research Site, Overland Park, Kansas
  - Octapharma Research Site, Louisville, Kentucky
  - Octapharma Research Site, White Marsh, Maryland
  - Octapharma Research Site, Kansas City, Missouri
  - Octapharma Research Site, Omaha, Nebraska
- Germany (2):
  - Octapharma Research Site, Leipzig
  - Octapharma Research Site, Munich
- Hungary (2):
  - Octapharma Research Site, Budapest
  - Octapharma Research Site, Debrecen
- Italy (3):
  - Octapharma Research Site, Napoli
  - Octapharma Research Site, Roma
  - Octapharma Research Site, Treviso
- Octapharma Research Site, Krakow, Poland
- Octapharma Research Site, Bratislava, Slovakia
- Ukraine (2):
  - Octapharma Research Site, Kyiv
  - Octapharma Research Site, Lviv

IPD SHARING:
Plan to Share IPD: No